CLINICAL TRIAL: NCT04289961
Title: A Research Protocol for Collection of Peripheral and Portal Vein Blood From Patients With Pancreatic Adenocarcinoma for Translational Research
Brief Title: PDAC Peripheral and Portal Vein Sampling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Juan Valle, Professor of Medical Oncology, The Christie NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18_DOG03-436
Record Dates: First submitted 2018-07-26; First posted 2020-02-28 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Circulating Tumour Cells (CTCs); CTC clusters; EUS-FNA; Portal Vein; Biomarkers

STUDY DESIGN:
Intervention Model Description: Prospective translational research study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Observational study of CTC microemboli in portal vein blood samples.
  Interventions: Diagnostic Test: Portal vein sampling

INTERVENTIONS:
Diagnostic Test: Portal vein sampling — During Endoscopic UltraSound guided-Fine Needle Aspitation (EUS-FNA) a curvilinear echoendoscope is advanced to the distal stomach or duodenal bulb to provide a window of access to a branch of the PV. After verifying venous flow by Doppler signal, a 19-gauge EUS-FNA needle is advanced transhepatically into the portal vein branch. With the needle in the portal vein, the stylet is removed and negative-pressure suction is applied to aspirate blood. A transhepatic approach for portal vein branch access is an absolute requirement of this technique in order to minimize the risk of bleeding. The puncture site is monitored under EUS for complications.

SUMMARY:
This is a research study in which bio-specimens (whole blood, plasma and serum from peripheral circulation and portal vein) will be collected from patients with pancreatic adenocarcinoma for translational research. These samples will be used for (but not limited to) identification and characterisation of blood-borne biomarkers at the genomic and protein expression level. Examples of such biomarkers are circulating tumour cells (CTCs), CTC clusters and circulating DNA (which can be tumour derived, or from unaffected/normal cells). CTC-enriched blood samples may also be used to generate CTC-derived tumour explant (CDX) models in immunocompromised mice in order to produce suitable disease models in which to test novel therapies and identify new molecular targets. In addition, permission will be sought from study participants for the research team to access clinical information from medical notes to aid in determining the clinical relevance of biomarkers identified during the course of this study. Validated biomarkers are anticipated to be used in designing future biomarker-directed clinical trials in these disease groups.

DETAILED DESCRIPTION:
Pancreatic Ductal Adenocarcinoma (PDAC) presents an urgent medical need. Approximately 9000 new cases of pancreatic cancer are diagnosed every year in the United Kingdom (UK) and worldwide it is projected to become the second most common cause of cancer related death by 2030. Currently the diagnostic pathway starts with pancreatic protocol Computed Tomgraphy (CT) scan which demonstrates sensitivity of 90% and specificity of 99% in diagnosis of pancreatic cancer. Magnetic Resonance Imaging (MRI) and Positron Emission Tomography (PET) can assist with ambiguous masses. Despite the high sensitivity and specificity of imaging modalities, definitive diagnosis is routinely obtained only by endoscopic ultrasound (EUS)-guided fine-needle aspiration (FNA). During this procedure four "passes" (biopsies) on average are required to obtain sufficient tissue for diagnosis.

Patients usually present with locally advanced or metastatic disease and are offered standard of care chemotherapy, which has only a limited impact on overall survival. Consequently the 5-year overall survival (OS) is only 2% with no significant improvement over the last 40 years. Approximately only 20% of the patients are eligible for surgical resection which is followed by adjuvant chemotherapy. However, 66% of these patients will experience local or distant recurrence, leading to a median overall survival in the range of 28 months. Improved stratification of patients for existing treatments may thus avoid unnecessary overtreatment and associated side effects to improve quality of life; conversely, it may also enable selection for a more appropriate treatment.

A significant reason for the lack of progress in tackling metastatic disease is the poor understanding of the biology and pathophysiology of metastasis. Studying the biology of PDAC metastasis is hampered by the fact that it is difficult to obtain tissue from the primary and metastatic sites. Moreover, serial biopsies following progression during treatment is largely not feasible, further hindering insight into the mechanisms of development of treatment resistance. The only easily-accessible blood-borne biomarker that is currently used in clinic is the serum marker carbohydrate antigen (CA) 19-9. However, its clinical use is limited firstly by the fact that 5-10% of the population are Lewis blood group negative and do not express CA19-9. Furthermore it is elevated in non-malignant pancreatic and extra-pancreatic diseases. Finally, CA19-9 cannot provide information about the genetic landscape that drives PDAC metastasis.

Metastatic spread is primarily haematogenous whereby tumour cells enter the circulation to metastasize mainly to the liver and lung. Such tumour cells have been shown to travel either as single circulating tumour cells (CTCs) or as groups of cells termed Circulating Tumour Microemboli (CTM). Heterogeneous CTM composed of cells expressing either epithellial or mesenchymal markers were isolated from patients with pancreatic cancer using a filtration-based method, the Isolation by Size of Epithelial Tumour cells platform (ISET), in a study performed at the Christie NHS Foundation Trust. As such, isolation and characterisation of CTCs and CTM will provide new insight into the underlying biological dependencies of metastasizing tumour cells and may thus provide opportunities to develop better and more accurate diagnostic and prognostic assays as well as opportunities to treat metastatic disease.

Detection and isolation of CTCs and CTM is limited by the fact that they represent very rare events compared to other cellular elements in the circulation. To this end, methods exploiting characteristics that differentiate CTCs from blood cells have been developed to overcome this obstacle. These CTC workflows usually start by enriching CTCs from a blood sample utilizing either surface markers present exclusively on CTCs, or their unique physical properties such as size, inertia, dielectric charge and density. Following enrichment, CTCs are isolated and can be simply enumerated or they are used for more advanced downstream analysis including genomic, transcriptomic and proteomic analysis as well as in vivo applications in cell culture and mouse models, with the aim of gaining insight into their function as metastatic seeds and biomarker development.

In the clinical setting, CTCs can be used to aid decision making. Indeed, enumeration of CTCs detected by the CellSearch platform has been FDA approved for prognosis and monitoring of metastatic breast, colorectal and prostate cancer. However, isolation and enumeration of CTCs in pancreatic cancer has given inconsistent results between studies as to whether CTCs can be used as prognostic biomarkers. These studies analysed CTCs isolated from peripheral blood. However, as the main venous drainage of the pancreas is through the portal vein to the liver, it may be hypothesized that CTCs could be filtered and removed as they pass through the liver capillaries. Hence, in order to define the biological and prognostic role of CTCs in pancreatic adenocarcinoma, it is critical to initiate studies with blood isolated from the portal vein to bypass confounding effects. Indeed, detection of CTCs in portal vein (PV) blood acquired at operation was recently reported by Bissolati et al.. By obtaining peripheral vein samples at the same time, this study confirmed that CTC number was greater in portal compared to peripheral samples and also demonstrated significant correlation between CTC positivity in portal vein samples and frequency on liver metastasis. However, it failed to show significant correlation with OS or Disease Free Survival (DFS). PV sampling has been performed safely; in December 2015 Catenacci et al. reported collection of PV blood from 18 patients with pancreatobilliary cancers by EUS-FNA with no complications during the procedure. PV puncture has also been previously reported for islet cell transplantation in patients with Type 1 Diabetes Mellitus. This procedure has low morbidity and also, potential complications, such as portal vein thrombosis, perihepatic or intraparenchymal hepatic haemorrhage and haemothorax are reported at a low rate.

During EUS-FNA a curvilinear echoendoscope is advanced to the distal stomach or duodenal bulb to provide a window of access to a branch of the PV. After verifying venous flow by Doppler signal, a 19-gauge EUS-FNA needle is advanced transhepatically into the portal vein branch. With the needle in the portal vein, the stylet is removed and negative-pressure suction is applied to aspirate blood. A transhepatic approach for portal vein branch access is an absolute requirement of this technique in order to minimize the risk of bleeding. The puncture site is monitored under EUS for complications. As tumour tissue will be obtained at the same time, a potential risk is the introduction of cancer cells into the circulation as the needle is withdrawn from the tumour. This risk however is circumvented as the route of the needle into the portal vein would avoid the primary mass.

The primary reason for drug failure in PDAC is the failure to identify predictive biomarkers for treatment response which would allow enrichment of patient sub-groups most likely to benefit from an individual therapy. This is in contrast to other major cancer types, in which advances in development of new cancer therapeutics and resulting improvement in survival outcomes are mainly due to the use of predictive biomarkers to select patients who will derive differential benefit from a particular therapeutic agent. Trastuzumab in breast cancers over-expressing HER-2, cetuximab for KRAS wild-type colorectal cancer, and gefitinib and erlotinib for Epidermal Growth Factor Receptor (EGFR) mutant non-small cell lung cancer best exemplify this therapeutic paradigm. By providing greater numbers of CTCs and CTM, analysis of PV sample will enable studies of their biology as well as development of cell lines and CDX models to allow identification of novel biomarkers and targets for new treatments.

Considering current gaps in knowledge of tumour biology of PDAC and the lack of progress in therapeutics, there is an urgent clinical need to develop a research strategy that will allow the discovery and validation of new biomarkers in this group of patients, and inform on biomarker-directed clinical trials to ultimately improve survival. To initiate such a research strategy, there is a need for systematic, prospective collection and analysis of blood samples acquired from peripheral and portal vein circulation to identify blood-borne surrogate tumour markers that will enable physicians to obtain relevant information for making personalised therapeutic decisions, in a minimally-invasive way.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically-suspected or cytologically/histologically-proven Pancreatic Adenocarcinoma who have been referred for EUS-FNA. Patients who are already on treatment would also be eligible.
2. Patients who are 18 years or older.
3. Patients must be able to receive and understand verbal and written information regarding the study and give written informed consent.
4. Patients must be able to comply with trial requirements.

Exclusion Criteria:

1. Patients with other active malignancy would not be eligible with the exception of patients with squamous or basal cell carcinoma of the skin. An exception to this statement would be those patients with a known/suspected germ-line predisposition to suffer multiple malignancies, such as, but not limited to Hereditary Breast and Ovarian Cancer Syndrome (BRCA1/2), Lynch syndrome or multiple endocrine neoplasia (MEN) syndrome.
2. Patient with INR >1.5 and/or platelets ≤50.
3. Patients with bleeding disorders.
4. Patients on anti-platelet or anti-coagulation treatment that cannot be temporarily discontinued around the procedure.
5. Patients who cannot give informed consent.
6. Patients with known Hepatitis C viral infection.
7. Patients with known Human Immunodeficiency Virus (HIV) infection.
8. If clinically judged by the investigator that the patient should not participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Blood-borne biomarker analysis for PDAC | 12 months
  To prospectively collect paired peripheral and portal vein serum, plasma and whole blood samples for translational research at various time points. To investigate the presence of Circulating Tumour Cells and Circulating Tumour Microemboli and their biological significance. To investigate potential prognostic and predictive blood-borne genetic, protein and/or messenger ribonucleic acid biomarkers using the collected specimens.

SECONDARY OUTCOMES:
Correlation of identified biomarkers with progression free and overall survival | 24 months
  To prospectively collect progression free and overall survival data so that correlation between biomarker parameters and clinical parameters can be examined.
Investigation germline genetic biomarkers | 12-24 months
  Investigation of potential predictive blood germline genetic biomarkers using the collected specimens.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Manchester University NHS Foundation Trust, Manchester
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No
Identifiable personal data (IPD) will be reviewed by the investigators listed on the trial delegation log at the stage of reviewing the medical records during the hepatopancreatobiliary (HPB) MultiDisciplinary Team (MDT) meeting at Manchester University Foundation Trust where the recruitment process will start. The medical notes will also be reviewed to correlate biomarker research with clinical outcomes. However, no participants' identifiable information will be shared with anyone outside the clinical or research team.